CLINICAL TRIAL: NCT02947360
Title: The FOVUS-ER Study: Focused Vascular Ultrasound to Risk Stratify Patients With Suspected Ischemic Chest Pain in the Emergency Department
Brief Title: The FOVUS-ER Study: Focused Vascular Ultrasound to Risk Stratify Patients With Chest Pain in the ER
Acronym: FOVUS-ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Steven Brooks, Associate Professor, Principal Investigator, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EMED-243-16
Record Dates: First submitted 2016-10-26; First posted 2016-10-27 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Carotid Artery Plaque
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOVUS (Experimental): All eligible and consenting patients will receive a focused vascular ultrasound examination of the carotid arteries
  Interventions: Other: Focused vascular ultrasound of the carotid arteries

INTERVENTIONS:
Other: Focused vascular ultrasound of the carotid arteries — Emergency physicians and a trained research sonographer will perform a focused vascular ultrasound of the carotids (FOVUS) in patients presenting to the emergency department with chest pain. The diagnostic test characteristics (sensitivity, sensitivity, negative predictive value, positive predictive value and likelihood ratios) for FOVUS carotid plaque height will be determined in relation to our primary outcome (30-day major adverse cardiac events)
  Other Names: FOVUS

SUMMARY:
Broad Goal: To demonstrate that focused vascular ultrasound (FOVUS) can accurately risk stratify patients with chest pain in the emergency department (ED).

Background and Rationale: Traditional risk assessment focuses on characteristics of the pain, known Coronary Artery Disease (CAD), risk factors, electrocardiogram (ECG), and blood tests to identify active ischemia. Identifying clinically significant CAD remains one of the most challenging tasks in the ED. Current clinical decision rules err on the side of over investigation and admission. To address this limitation, the Investigators have developed a point-of-care carotid ultrasound test predictive of CAD. The Investigators have shown that carotid plaque is strongly associated with significant angiographic CAD in a population referred for angiogram.

Research Aims:

Primary - To determine the association between carotid plaque measured by a dedicated sonographer and 30-day major adverse cardiac events (MACE), including MI, reperfusion, or death in patients presenting to the ED with suspected cardiac ischemia.

Secondary - To determine the agreement sonographer and emergency physician FOVUS results.

Methodology: The Investigators propose a prospective cohort study to assess the prognostic value of a novel point-of-care carotid ultrasound plaque quantification protocol in the ED of Kingston General Hospital. We will enroll 500 consecutive patients presenting with a chief complaint of chest pain prompting at least one 12-lead ECG and troponin measurement. Patients will undergo carotid scan by a dedicated sonographer and emergency physician. Patients will be followed for MACE for 30 days. Those performing scans will be blinded to clinician's impression and care plans while clinicians will be blinded to FOVUS findings. The primary analysis will involve determination of the sensitivity, sensitivity, positive predictive value, negative predictive value and likelihood ratios associated with FOVUS for 30-day MACE.

Expected Outcomes: The study will provide evidence to determine whether FOVUS may be a useful prognostic tool for emergency physicians assessing patients with suspected ischemic chest pain. The secondary analysis will provide evidence to determine whether emergency physicians can be trained to measure carotid plaque height accurately when compared to the gold standard ultrasonographer measurement.

Significance: If FOVUS can reliably identify very low risk patients, implementation of this novel tool could reduce ED length of stay, monitoring, and overcrowding.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥25 years of age;
2. Chief complaint of chest pain possibly due to coronary ischemia and requiring cardiac investigations (e.g. ECG, troponin) in the opinion of the treating emergency physician;
3. Receiving at least one 12-lead ECG;
4. Receiving at least one serum troponin measurement;
5. Willing to provide informed consent.

Exclusion Criteria:

1. Acute ST-segment elevation on the initial ECG;
2. Hemodynamic instability;
3. High clinical suspicion of pulmonary edema;
4. History of recent cocaine or amphetamine use;
5. Inability to communicate in English;
6. A clear traumatic etiology;
7. Prior enrollment in the study within the past 6 months;
8. Terminal non-cardiac illness;
9. Previous carotid surgery (endarterectomy or stent);
10. Anatomic consideration rendering carotid artery inaccessible (tumor, abscess, scarring, mechanical device).

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 30 days
  Major adverse cardiac events will include acute myocardial infarction (MI),revascularization or mortality

SECONDARY OUTCOMES:
Plaque height measurement during FOVUS | At enrollment
  Agreement between ultrasonographers and emergency physicians with respect to plaque height measurement will be calculated using this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Brooks, MD, MHSc, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brooks SC, Sivilotti MLA, Hetu MF, Norman PA, Day AG, O'Callaghan N, Latiu V, Newbigging J, Hill B, Johri AM. Focused carotid ultrasound to predict major adverse cardiac events among emergency department patients with chest pain. CJEM. 2023 Jan;25(1):81-89. doi: 10.1007/s43678-022-00395-w. Epub 2022 Oct 31. PMID 36315347